CLINICAL TRIAL: NCT05205044
Title: Evaluation of Apelin-13 and Apelin-36 Concentrations in Women With Primary Unexplained Recurrent Pregnancy Loss
Brief Title: Evaluation of Apelin-13 and Apelin-36 in Women With Recurrent Pregnancy Loss
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MS 672/2021
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Recurrent Pregnancy Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent pregnancy loss
  Interventions: Diagnostic Test: Apelin-13, Apelin-36
- Healthy
  Interventions: Diagnostic Test: Apelin-13, Apelin-36

INTERVENTIONS:
Diagnostic Test: Apelin-13, Apelin-36 — Serum levels of Apelin-13 and Apelin-36

SUMMARY:
Lower Apelin levels are associated with hypertensive disorders with pregnancy, yet no studies investigated its levels in recurrent pregnancy loss

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in first trimester
* negative antiphospholipid markers
* normal karyotype

Exclusion Criteria:

* multiple pregnancy
* fetal malformations
* maternal diseases
* smoking or alcohol use
* history of or risk factors for preterm labor

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant females in first trimester
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2022-01-23 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Apelin-13 and Apelin-36 | 1 year
  Serum levels of Apelin-13 and Apelin-36

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain Shams University Maternity Hospital, Cairo, Cairo/القاهرة
  - AinShams Maternity Hospital, Cairo

IPD SHARING:
Plan to Share IPD: Undecided